CLINICAL TRIAL: NCT00004863
Title: A Phase I Open-Label Safety Study of Escalating Doses of Taxol in Combination With Escalating Doses of GEM231 in Patients With Refractory Solid Tumors
Brief Title: Paclitaxel and GEM 231 in Treating Patients With Recurrent or Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000067518; P30CA013330 (NIH); AECM-1199906196; HYBRIDON-231-100B; NCI-G00-1665
Record Dates: First submitted 2000-03-07; First posted 2004-03-15 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — GEM231; Paclitaxel

INTERVENTIONS:
Drug: GEM 231
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of paclitaxel and GEM 231 in treating patients who have recurrent or refractory solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety and maximum tolerated dose of GEM 231 and paclitaxel in patients with recurrent or refractory solid tumors. II. Determine any preliminary antitumor activity of this regimen in these patients.

OUTLINE: This is a dose escalation study of GEM 231. Patients receive paclitaxel IV over 3 hours on day 1, immediately followed by GEM 231 over 2 hours on days 1, 4, 8, 11, 15, and 18. Treatment continues every 3 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients are treated with one of two doses of paclitaxel and escalating doses of GEM 231 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which no more than 2 of 6 patients experience dose limiting toxicity. Patients are followed monthly for 3 months.

PROJECTED ACCRUAL: A maximum of 1 patient will be accrued per week for this study until the maximum tolerated dose is reached.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed advanced solid tumor that is refractory to standard therapy or for which no standard therapy exists Measurable or evaluable disease No CNS metastases that are untreated, associated with seizures, or require intravenous medication and/or hospitalization

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: WHO 0-2 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 8.5 g/dL Hepatic: Bilirubin no greater than upper limit of normal (ULN), except with Gilbert's syndrome (no greater than 1.5 times ULN if liver metastases present) PT and aPTT normal SGOT or SGPT less than 3 times ULN (no greater than 5 times ULN if liver metastases present) Renal: Creatinine less than 1.25 times ULN No renal tubular dysfunction (i.e., at least 2+ proteinuria within the past 2 weeks) Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception for 1 month prior to, during, and 3 months after study No other serious medical condition that would prevent compliance No serious infection No known hypersensitivity to paclitaxel or other drugs formulated in Cremophor or any oligodeoxynucleotides Adequate venous access No psychological or geographical condition that would prevent compliance

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 1 week since prior transfusion Prior biologic therapy allowed and recovered No concurrent biologic therapy Chemotherapy: Prior chemotherapy allowed and recovered No other concurrent chemotherapy Endocrine therapy: Prior hormonal therapy allowed and recovered Concurrent palliative hormonal therapy allowed Radiotherapy: Prior radiotherapy allowed and recovered No concurrent radiotherapy (except palliative) Surgery: At least 2 weeks since prior major surgery with wound complications Other: At least 2 weeks since prior investigational drugs No other investigational drugs during or within 28 days of study No concurrent CYP-3A metabolism dependent drugs

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 1999-07 (Actual); Primary Completion 2001-08 (Actual); Study Completion 2001-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sridhar Mani, MD, Study Chair — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein Comprehensive Cancer Center, The Bronx, New York, United States